CLINICAL TRIAL: NCT04618224
Title: Introduction of an Internet-based Near and Intermediate-vision Reading Test for Greek-speaking Normal and Low Vision Adults (wDDART): Development and Validation.
Brief Title: Development and Validation of an Internet-based Near and Intermediate-vision Reading Test
Acronym: wDDART
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES13/Th29/22-10-2020
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Presbyopia; Refractive Errors; Low Vision; Near Vision; Reading
Keywords: internet-based digital reading test; smart features; face detection; reading acuity; reading speed; critical print size
MeSH Terms: conditions — Presbyopia; Refractive Errors; Vision, Low; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: * 70 patients with normal vision (NVG) with adequate literacy of written Greek language
  * 30 patients with low vision (LVG) with adequate literacy of written Greek language
  These patients are tested on the digital reading test DDART.
  Interventions: Diagnostic Test: DDART Testing
- Study group: The same patients as those in the control group (NVG, LVG) are tested on the online version of the Greek digital reading test DDART (wDDART).
  Interventions: Diagnostic Test: wDDART Testing

INTERVENTIONS:
Diagnostic Test: DDART Testing — One randomly selected eye is included for each study participant. Participants respond to the DDART near vision test with defined environmental conditions at 40 cm viewing distance. All four parameters (RA, MRS, CPS and ACC) are evaluated.
  Groups: Control group
Diagnostic Test: wDDART Testing — One randomly selected eye is included for each study participant. Participants respond to the wDDART near vision test with defined environmental conditions at 40 cm viewing distance. All four parameters (RA, MRS, CPS and ACC) are evaluated.
  Groups: Study group

SUMMARY:
Primary objective of our study is to develop and validate an internet-based digital near and intermediate-vision reading test in the greek language.

DETAILED DESCRIPTION:
Present study aims to develop and validate a computer-based digital near-vision reading test (web Democritus Digital Acuity Reading Test - wDDART) based on the validated digital DDART.

Specifically, present study aims to develop a new online reading test (wDDART) based on the corresponding digital DDART reading test for Windows and to evaluate the level of agreement between the two reading tests, as well as test-retest reliability of the online wDDART reading test.

The first part of the study is the development of the online reading test, which will include the following new smart features:

1. Automatic calculation of the reading time of each sentence (each logMAR)
2. Automatic calculation of the basic reading parameters - RA, MRS, CPS, ACC - immediately after the completion of the examination
3. Adjustment of the font size according to the size of the computer screen used for the examination
4. Real time calculation of the patient-screen distance through a face detection system

The second part of this study is the clinical validation of the online wDDART reading test. In this part, four reading parameters measured with the digital and the online version are compared. These parameters are the following:

1. Reading Acuity (RA)
2. Maximum Reading Speed (MRS)
3. Critical Print Size (CPS)
4. Accessibility Index (ACC) All the comparisons take place in two groups: a) a Normal Vision Group (NVG), and b) a Low Vision Group (LVG) in order to estimate the reading capacity in a population with a wide range of vision.

ELIGIBILITY:
Inclusion Criteria:

* Adequate literacy of written Greek language
* Age between 18 to 75 years

Exclusion Criteria:

* Dyslexia
* Attention-deficiency
* Former diagnosis of mental and/or psychiatric diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal- and low-sighted participants aged 18 to 75 years
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Reading Acuity (RA) | through study completion, an average of 3 months
  The smallest print that can be read by the patient easily (measured in logMAR). It is calculated by the following formula:
  RA = 1.4 - (sentences x 0.1) + (errors x 0.01).
Maximum Reading Speed (MRS) | through study completion, an average of 3 months
  The patient's reading speed (measured in wpm) when reading is not limited by print size. It is calculated by averaging the reading speed of the sentences with print size larger than the CPS.
Critical Print Size (CPS) | through study completion, an average of 3 months
  The smallest print size (measured in logMAR) that can be read with the MRS, i.e., with speed greater than or equal to the average reading speed of the larger logMAR print sentences minus 1.96 times the standard deviation (SD) of the reading speed of these sentences.
Accessibility Index (ACC) | through study completion, an average of 3 months
  The mean reading speed of the 10 largest print sizes at 40 cm (1.3 to 0.4 logMAR), divided by 200 wpm, which is the mean reading speed of normally sighted young adults aged 18 to 39 years old. This parameter was designed for better evaluation of one's access to text across the range of the 10 most common print sizes found in everyday life. For instance, a value of 0 means no access to commonly encountered printed material, while 1.0 is the mean value for normally sighted young adults that indicates reading fluency within the everyday life print sizes.

SECONDARY OUTCOMES:
Intraclass Correlation Coefficients (ICCs) for study participants | through study completion, an average of 3 months
  Level of agreement between the digital and the online version are evaluated by calculation of the ICCs for the 4 reading parameters (RA, MRS, CPS, ACC).

OTHER OUTCOMES:
Test-retest Intraclass Correlation Coefficients (ICCs) | through study completion, an average of 3 months
  Test-retest reliability of the internet-based reading test wDDART is evaluated by ICCs for the 4 reading parameters (RA, MRS, CPS, ACC).

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (2):
- Greece (2):
  - Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - Department of Computer Science and Biomedical Informatics, University of Thessaly, Lamía, Thessaly

REFERENCES:
- [Result] Labiris G, Panagiotopoulou EK, Chatzimichael E, Tzinava M, Mataftsi A, Delibasis K. Introduction of a digital near-vision reading test for normal and low vision adults: development and validation. Eye Vis (Lond). 2020 Oct 22;7:51. doi: 10.1186/s40662-020-00216-0. eCollection 2020. PMID 33102611
- [Derived] Labiris G, Panagiotopoulou EK, Duzha E, Tzinava M, Perente A, Konstantinidis A, Delibasis K. Development and Validation of a Web-Based Reading Test for Normal and Low Vision Patients. Clin Ophthalmol. 2021 Sep 22;15:3915-3929. doi: 10.2147/OPTH.S314943. eCollection 2021. PMID 34588763